CLINICAL TRIAL: NCT03742882
Title: A Phase 1, Open-label, Multicenter, Single-dose Study to Assess the Pharmacokinetics of CC-90001 in Subjects With Mild, Moderate, and Severe Hepatic Impairment Compared With Healthy Subjects
Brief Title: A Study to Assess the Pharmacokinetics of CC-90001 in Subjects With Mild, Moderate, and Severe Hepatic Impairment Compared With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90001-CP-005; U1111-1223-7431 (Other: WHO)
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Hepatic Impairment
Keywords: CC-90001; Pharmacokinetics; Hepatic Impairment; Healthy subjects
MeSH Terms: interventions — CC-90001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-90001 (Experimental): Single oral dose of 200 mg of CC-90001
  Interventions: Drug: CC-90001

INTERVENTIONS:
Drug: CC-90001 — CC-90001

SUMMARY:
This is a multicenter, open-label study to assess the PK of a single 200 mg oral dose of CC-90001 in subjects with mild, moderate, and severe hepatic impairment, and in matched healthy control subjects with normal hepatic function.

Degrees of hepatic impairment will be determined during screening by the subject's score according to Child-Pugh Classification Criteria.

DETAILED DESCRIPTION:
Subjects will be enrolled in Groups 1 through 5 as follows:

* Group 1: Approximately 6 to 8 male or female subjects with mild hepatic impairment (with a Child-Pugh score of ≥ 5 to ≤ 6) will be enrolled in Group 1.
* Group 2: Approximately 6 to 8 male or female subjects with moderate hepatic impairment (with a Child-Pugh score of ≥ 7 to ≤ 9) will be enrolled in Group 2.
* Group 3: Approximately 6 to 8 healthy male or female subjects with normal hepatic function will be enrolled in Group 3. Subjects in Group 3 will be matched to subjects in Group 2 with respect to sex, age (± 10 years), and weight (± 10% body mass index [BMI]). Group 3 will also serve as the control group for Group 1.
* Group 4: Approximately 6 to 8 male or female subjects with severe hepatic impairment (with a Child-Pugh score of ≥ 10 to ≤ 13) will be enrolled in Group 4.
* Group 5: Approximately 6 to 8 healthy male or female subjects with normal hepatic function will be enrolled in Group 5. Subjects in Group 5 will be matched to subjects in Group 4 with respect to sex, age (± 10 years), and weight (± 10% BMI).

This study employs a staged design as follows:

* Subjects with mild or moderate hepatic impairment and matching healthy subjects with normal hepatic function (Groups 1 through 3) will be enrolled concomitantly.
* At least 4 subjects with mild or moderate hepatic impairment must demonstrate satisfactory safety and tolerability for up to 4 days after dosing before subjects with severe hepatic impairment may be dosed.
* Two subjects with severe hepatic impairment must demonstrate satisfactory safety and tolerability for up to 4 days after dosing before the remaining subjects with severe hepatic impairment may be dosed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements, including the restrictions.
3. Subject is male, or non-pregnant and non-nursing female between ≥ 18 and ≤ 70 years of age at the time of signing the ICF.
4. Subject has Body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at screening.
5. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle-stimulating hormone [FSH] level in the postmenopausal range according to the laboratory used at Screening); FSH to be performed at the discretion of the Investigator in consultation with the Medical Monitor.
6. Females of childbearing potential (FCBP)1 must have a negative pregnancy test at the Screening and Baseline Visits. While receiving Investigational Product (IP) and for at least 28 days after taking the dose of IP, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below: Option 1: One highly effective method (e.g., hormonal contraception [oral, injection, implant, transdermal patch, vaginal ring]; intrauterine device; tubal ligation; or partner's vasectomy) and one additional form (latex condom or any nonlatex condom not made of natural [animal] membrane [eg, polyurethane], diaphragm, sponge).

   OR Option 2: Male or female condom PLUS 1 additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
7. Male subjects must:

   a. Practice true abstinence2 (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms were recommended]) during sexual contact with a pregnant female or female of FCBP while participating in the study, during dose interruptions, and for at least 28 days after the dose of investigational product, even if he has undergone a successful vasectomy.
8. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator.
9. Subject is afebrile (febrile is defined as ≥ 38°C or 100.3°F), with supine systolic blood pressure ≥ 90 and ≤ 160 mm Hg, supine diastolic blood pressure ≥ 50 and ≤ 100 mm Hg, and pulse rate ≥ 40 and ≤ 100 beats per minute at Screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study at the Investigator's discretion.
2. Subject has any condition that places the subject at an unacceptable risk if he or she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject is pregnant or breastfeeding.
5. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever was longer).
6. Subject has used moderate or strong CYP3A4/5 inducers and/or inhibitors (including St. John's wort) within 30 days prior to dosing. The Indiana University P450 Drug Interactions Flockhart Table™ may be consulted for a list of such medications (http://medicine.iupui.edu/clinpharm/ddis/main-table).
7. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. Subjects with appendectomy and cholecystectomy may be included.
8. Subject has an estimated creatinine clearance < 60 mL/min as calculated using the Cockcroft-Gault formula.
9. Subject has donated blood or plasma within 2 weeks before dose administration to a blood bank or blood donation center.
10. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs unless positive drug screen is due to prescription drug use that is approved by the Investigator and the Medical Monitor.
11. Subject has a history of alcohol abuse (as defined by the current version of the Diagnostic and Statistical Manual) within 1 year before dose administration, or a positive alcohol screen.
12. Subject has had a positive result to the test for human immunodeficiency virus (HIV) antibodies at Screening.

    • Chronic or resolved Hepatitis B or Hepatitis C are acceptable only if sequelae are limited to hepatic involvement and its consequent comorbidities. (ie, vasculitis, clinically significant globulinemia, etc. are unacceptable).
13. Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
14. Subject has received live vaccination (excluding seasonal flu vaccination) within 30 days of dosing.
15. Subject is part of the clinical staff personnel or a family member of the study site staff.
16. Subject is, for any reason, deemed by the investigator to be inappropriate for this study, including a subject who is unable to communicate or to cooperate with the investigator or the clinical staff.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- AUC0-t | UP to approximately 7 Days
  Estimation of AUC calculated from time zero to the last measured time point
Pharmacokinetic- AUC0-∞ | UP to approximately 7 Days
  Estimation of AUC calculated from time zero to infinity
Pharmacokinetic- Cmax | UP to approximately Day 1
  Estimation of observed maximum plasma concentration
Pharmacokinetic- Tmax | UP to approximately Day 1
  Estimation of time to Cmax
Pharmacokinetic- t1/2 | Up to approximately 7 days
  Estimation of terminal elimination half-life
Pharmacokinetic- CL/F | Up to approximately 7 days
  Estimation of apparent clearance of drug from plasma after extravascular administration
Pharmacokinetic- Vz/F | Up to approximately 7 days
  Estimation of apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of subjects with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Kofi Mensah, MD, PhD, Study Director — Celgene
Locations (4):
- United States (4):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee
  - The Texas Liver Institute, San Antonio, Texas